CLINICAL TRIAL: NCT04856306
Title: Myomectomy vs Uterine Artery Embolization vs GnRh Antagonist for AUB-L
Acronym: Magical
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00002872
Record Dates: First submitted 2021-04-20; First posted 2021-04-23 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Heavy Menstrual Bleeding; Fibroid Uterus
Keywords: fibroids
MeSH Terms: conditions — Menorrhagia; Leiomyoma | interventions — Uterine Artery Embolization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Myomectomy: After routine patient counseling on fibroid treatments, this group chooses surgical myomectomy of any type (abdominal/laparoscopic/hysteroscopic)
  Interventions: Other: Groups 1 and 2 myomectomy and uterine artery embolization, respectively, are surgical/procedure
- Uterine artery embolization: After routine patient counseling on fibroid treatments, this group chooses uterine artery embolization procedure.
  Interventions: Other: Groups 1 and 2 myomectomy and uterine artery embolization, respectively, are surgical/procedure
- Elagolix: After routine patient counseling on fibroid treatments, this group chooses the following medication: every morning (AM), 300mg elagolix, 1mg estradiol, and 0.5mg norethindrone acetate capsules taken in one combined capsule and every evening (PM), 300mg elagolix capsule. In our study, this medication will be administered for 12 months unless the subject withdraws from the study. It is FDA-approved for continuous use of up to 24 months.
  Interventions: Drug: Elagolix Oral Product

INTERVENTIONS:
Other: Groups 1 and 2 myomectomy and uterine artery embolization, respectively, are surgical/procedure — See previous descriptions
  Groups: Myomectomy; Uterine artery embolization
Drug: Elagolix Oral Product — See group 3 description
  Other Names: Oriahnn
  Groups: Elagolix

SUMMARY:
This is a prospective cohort study comparing the novel FDA-approved oral GnRH antagonist ORIAHNN (elagolix, estradiol, and norethindrone acetate capsules; elagolix capsules) to uterine artery embolization (UAE) or myomectomy (abdominal, laparoscopic, or hysteroscopic) for treatment of heavy menstrual bleeding due to leiomyomas. Uterine leiomyomas, also called fibroids, are hormone-dependent growths in the uterine muscle that are common in reproductive-age women (1). Leiomyomas can often lead to heavy menstrual bleeding. Definitive treatment for abnormal uterine bleeding due to leiomyomas is hysterectomy, but for patients who desire uterine conservation, a variety of treatment options exist. Regulation of menses with combined oral contraceptives or progestin only oral formulations are generally considered first line treatment but are not curative or effective for many patients. Another treatment option is a myomectomy, which is the surgical resection or removal of myomas. Myomectomy can be performed via hysteroscopy or laparoscopy, or by a vaginal or an abdominal approach. The route of removal depends on myoma location and patient symptoms. Another treatment option is Uterine fibroid or uterine artery embolization (UFE/UAE). UAE is a minimally invasive procedure where permanent particles are delivered to and block/embolize the blood supply to the myoma via a fluoroscopy directed arterial catheter. This typically leads to a decrease in fibroid size and associated bleeding (2). ORIAHNN, an oral GnRH antagonist that was FDA-approved in 2020, has demonstrated significant decrease in myoma-associated heavy menstrual bleeding compared to placebo (1) but has not been compared to other standard of care interventions. The primary objective of this study is to compare this novel medication to the common AUB-L treatments UAE and Myomectomy.

DETAILED DESCRIPTION:
Uterine fibroids, or leiomyomas, are common benign tumors in reproductive-age women. While many women with fibroids are asymptomatic, 20-50% of women may have bulk symptoms, such as pelvic pressure, urinary or gastrointestinal symptoms, and/or heavy menstrual bleeding (3-4). Heavy menstrual bleeding can lead to severe anemia requiring treatment, which has negative health and economic consequences (4). Fibroids are also associated with infertility and recurrent pregnancy loss (3). Symptom character and severity depend on fibroid size and location, and they can have a significant effect on women's quality of life.

Fibroid growth is dependent on estrogen and progesterone, thus common medical management of symptoms uses hormonal agents, such as oral contraceptives, selective progesterone receptor modulators, GnRH agonists, and intrauterine devices (3). Nonhormonal medical methods include tranexamic acid, an antifibrinolytic agent that reduces menstrual blood loss, and nonsteroidal anti-inflammatory drugs, which reduce blood loss and improve pain relief (3). Medical management is generally the first treatment strategy for symptomatic fibroids, but definitive treatment is via a hysterectomy. A hysterectomy is the most common surgical treatment of fibroids, but for women who desire to preserve the uterus, other surgical options are available (4, 5). A myomectomy removes fibroids employing either hysteroscopic, laparoscopic, abdominal approaches, or a combination of these methods. Another option for fibroid management is uterine fibroid or uterine artery embolization (UFE/UAE). This minimally invasive procedure uses a catheter to inject permanent particles inside uterine arteries to occlude the blood supply to the fibroid(s). Both myomectomy and UAE have high patient satisfaction rates. Both modalities also carry the risk of necessitating future interventions if symptoms are not controlled or if fibroids recur (5). Patients who undergo UAE have a slightly higher risk of further interventions compared to myomectomy (5).

For women who do not desire any type of surgical intervention or the UAE procedure, a new type of medical treatment has become available. Oriahnn, produced by AbbVie, is a combination of elagolix, an oral nonpeptide GnRH antagonist, and add-back therapy with estradiol and norethindrone (1, 4). It is administered at a total daily dose of 600mg: 300mg elagolix with add-back therapy in the morning and 300mg elagolix alone at night (4). Elagolix results in rapid, reversible suppression of gonadotrophin and ovarian sex hormones, and was first approved for treatment of endometriosis-associated pain (4). The side effects of elagolix are related to the creation of the hypoestrogenic state and are mitigated with add-back therapy (4). The dose and formula in Oriahnn showed a significant decrease in menstrual blood loss compared to placebo with a favorable safety profile but has never been compared to any other treatment for fibroids (4). It is FDA-approved for a treatment duration of 24 months (1).

ELIGIBILITY:
Inclusion Criteria:

Patients with heavy menstrual bleeding and uterine fibroids documented on imaging who are seeking treatment, and after completing standard counseling, chose either ORIAHNN, UAE, or myomectomy. If the patient has used hormonal treatments for fibroids in the past, a wash-out period of at least 3 months duration must be performed prior to study participation. If the patient has had a myomectomy of any type in the past, a period of at least 6 months must have passed since the surgery prior to study participation.

Exclusion Criteria:

pregnancy, presence of persistent (defined as present on 2 or more consecutive ultrasounds) or complex ovarian cyst, active cancer, history of osteoporosis, current pelvic inflammatory disease, history of liver or renal failure, presence of coagulopathy that is unable to be corrected, or untreated thyroid disease, and having previously been treated with UAE, GnRH antagonist, or myomectomy within the past 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women being treated for heavy menstrual bleeding due to fibroids at a MedStar facility.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Menstrual blood loss | 12 months
  Raw values and quantitative change in menstrual blood loss per month from patient's baseline

SECONDARY OUTCOMES:
UFS-QOL Score | 12 months
  Raw score and change in overall health-related quality of life score from UFS-QOL from patient's baseline at 3, 6, and 12-month intervals
Menopausal symptoms | 12 months
  Raw score and change in overall menopausal symptoms score based on Menopausal Symptoms questionnaire from patient's baseline at 3, 6, and 12-month intervals
Hemoglobin value | 12 months
  Hemoglobin laboratory values collected prior to treatment initiation and at 3-, 6-, 9-, and 12-month intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Hazen, MD, Study Director — MedStar Health; James Robinson, MD, Study Director — MedStar Health
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schirf BE, Vogelzang RL, Chrisman HB. Complications of uterine fibroid embolization. Semin Intervent Radiol. 2006 Jun;23(2):143-9. doi: 10.1055/s-2006-941444. PMID 21326757
- [Background] De La Cruz MS, Buchanan EM. Uterine Fibroids: Diagnosis and Treatment. Am Fam Physician. 2017 Jan 15;95(2):100-107. PMID 28084714
- [Background] Spies JB, Coyne K, Guaou Guaou N, Boyle D, Skyrnarz-Murphy K, Gonzalves SM. The UFS-QOL, a new disease-specific symptom and health-related quality of life questionnaire for leiomyomata. Obstet Gynecol. 2002 Feb;99(2):290-300. doi: 10.1016/s0029-7844(01)01702-1. PMID 11814511
- [Background] Gupta JK, Sinha A, Lumsden MA, Hickey M. Uterine artery embolization for symptomatic uterine fibroids. Cochrane Database Syst Rev. 2014 Dec 26;2014(12):CD005073. doi: 10.1002/14651858.CD005073.pub4. PMID 25541260
- [Background] Goodwin SC, Bradley LD, Lipman JC, Stewart EA, Nosher JL, Sterling KM, Barth MH, Siskin GP, Shlansky-Goldberg RD; UAE versus Myomectomy Study Group. Uterine artery embolization versus myomectomy: a multicenter comparative study. Fertil Steril. 2006 Jan;85(1):14-21. doi: 10.1016/j.fertnstert.2005.05.074. PMID 16412720
- [Background] Wyatt KM, Dimmock PW, Walker TJ, O'Brien PM. Determination of total menstrual blood loss. Fertil Steril. 2001 Jul;76(1):125-31. doi: 10.1016/s0015-0282(01)01847-7. PMID 11438330
- [Background] Magnay JL, Nevatte TM, O'Brien S, Gerlinger C, Seitz C. Validation of a new menstrual pictogram (superabsorbent polymer-c version) for use with ultraslim towels that contain superabsorbent polymers. Fertil Steril. 2014 Feb;101(2):515-22. doi: 10.1016/j.fertnstert.2013.10.051. Epub 2013 Dec 12. PMID 24331833
- [Background] Larsen L, Coyne K, Chwalisz K. Validation of the menstrual pictogram in women with leiomyomata associated with heavy menstrual bleeding. Reprod Sci. 2013 Jun;20(6):680-7. doi: 10.1177/1933719112463252. Epub 2012 Nov 27. PMID 23188490
- [Result] Schlaff WD, Ackerman RT, Al-Hendy A, Archer DF, Barnhart KT, Bradley LD, Carr BR, Feinberg EC, Hurtado SM, Kim J, Liu R, Mabey RG Jr, Owens CD, Poindexter A, Puscheck EE, Rodriguez-Ginorio H, Simon JA, Soliman AM, Stewart EA, Watts NB, Muneyyirci-Delale O. Elagolix for Heavy Menstrual Bleeding in Women with Uterine Fibroids. N Engl J Med. 2020 Jan 23;382(4):328-340. doi: 10.1056/NEJMoa1904351. PMID 31971678
- [Result] Broder MS, Goodwin S, Chen G, Tang LJ, Costantino MM, Nguyen MH, Yegul TN, Erberich H. Comparison of long-term outcomes of myomectomy and uterine artery embolization. Obstet Gynecol. 2002 Nov;100(5 Pt 1):864-8. doi: 10.1016/s0029-7844(02)02182-8. PMID 12423842
- See also: 1. FDA Approves the First Oral Medication for the Management of Heavy Menstrual Bleeding Due to Uterine Fibroids in Pre-menopausal Women AbbVie Press Release. May 29, 2020. — https://news.abbvie.com/news/press-releases/fda-approves-first-oral-medication-for-management-heavy-menstrual-bleeding-due-to-uterine-fibroids-in-pre-menopausal-women.htm